CLINICAL TRIAL: NCT06330779
Title: Trauma-adapted Yoga in Child & Adolescent Psychiatry: a Multicenter Study.
Brief Title: Trauma-adapted Yoga in Child & Adolescent Psychiatry.
Acronym: TAY-CAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University West, Sweden (Other)
Collaborators: Vastra Gotaland Region (Other Government); Healthcare Region Dalarna (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UWest
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: ADHD; PTSD; Quality of Life; Self-Control; Pain; Affect
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Stress Disorders, Post-Traumatic; Self-Control; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga-group (Experimental): 8 weeks ,once a week, instructor led trauma-adapted yoga intervention.
  Interventions: Other: Trauma-adapted yoga
- Controll (No Intervention): Waiting list

INTERVENTIONS:
Other: Trauma-adapted yoga — Trauma-adapted-yoga (TAY) classes The classes, which span eight weeks with a once-a-week frequency, each last approximately 45-50 minutes. These small group classes are structured in a semi-circle arrangement to create a sense of security and empowerment for the participants. The teaching approach is trauma-sensitive, characterized by its inviting nature, provision of choices when facing challenges (A-B choices), and direction toward tangible physical sensations to enhance interoceptive awareness. Each yoga session follows a structured sequence of activities designed to promote participants' well-being and physiological awareness.
  Online TAY classes After eight weeks, adolescents in the yoga group can continue their practice online. Exclusive to previous in-person participants, they'll receive a link for recorded classes and they will have the possibility to contact their health care contact any time.
  Arms: Yoga-group

SUMMARY:
The goal of this randomized clinical trial is to evaluate the efficacy of trauma-adapted yoga as a complementary intervention to care as usual in child and adolescents psychiatry clinics, in the population of adolescents with the diagnosis of ADHD and/or PTSD. We hypothesize that trauma-adapted yoga (TAY) is an effective non-pharmacological intervention for adolescent with ADHD and/or PTSD. Aims: (1) Validate the impact of TAY on the mental health & quality of life of adolescents with ADHD and/or PTSD. (2) Investigate the feasibility of online TAY for continued self-care. (3) Explore adolescents' experiences & parental perspectives on TAY in their treatment. (4) Explore healthcare professionals' experience on the integration of TAY into clinical practice.

Within and between group (yoga group vs waiting list) analyses will be performed.

DETAILED DESCRIPTION:
Study Summary

Introduction:

There is growing interest in applying yoga and mindfulness techniques to children and adolescents, although research in this area remains limited. Existing studies suggest that yoga can reduce stress, improve mood, enhance resilience, and boost self-regulation skills in school settings. Additionally, these approaches hold promise for improving mental health in clinical child and adolescent populations.

Study Aim:

The aim of this study is to evaluate the impact of trauma-adapted yoga (TAY) as a complement to care as usual in Child and Adolescent Psychiatry (CAP) clinics in the USA and Sweden. The study hypothesizes that eight weeks of TAY practice will reduce negative affect states and pain intensity/frequency, while improving emotional and behavioral control, attention, and resilience. It is expected that TAY will enhance the success of other ongoing treatments in CAP, foster improved well-being, and provide patients with self-care tools.

Importance of the Study:

The study's results are crucial for developing evidence-based care for children and adolescents with mental disorders and filling gaps in knowledge about yoga's efficacy as a treatment method.

Participants:

Adolescents aged 12-18 in contact with CAP clinics who have received a diagnosis of PTSD and/or ADHD are eligible. Inclusion criteria include understanding English or Swedish, while exclusion criteria involve ongoing substance use, active manic periods, psychotic disorders, suicidality, cognitive impairment, and serious physical illnesses.

Study Design:

The study adopts a Randomized Control Trial (RCT) design. Participants undergo pre-intervention assessment, followed by random assignment to either the yoga group or a control group. The yoga group attends weekly TAY sessions for eight weeks, while the control group waits. Assessments are conducted post-intervention and at a follow-up point. The study aims to include 174-180 adolescents.

Intervention:

TAY classes span eight weeks, incorporating physical movements, balance exercises, adapted breathing practices, trauma-informed mindfulness guidance, and guided progressive muscle relaxation. Participants have the option to continue yoga practice online after the intervention.

Assessment:

Assessment includes self-reported measures using validated instruments, such as the Child PTSD Symptom Scale, Positive/Negative Affect, Pain assessment, Child and Youth Resilience Measure, and Self-Directedness. Guardian-reported measures include the SNAP-IV and PedsQL-Fam inventory. Patient records provide additional data.

Qualitative Component:

After the intervention, individual interviews gather qualitative information on participants', guardians', and staff's experiences of yoga and its health effects.

This study aims to provide valuable insights into the potential benefits of trauma-adapted yoga for adolescents in CAP clinics, contributing to the advancement of evidence-based care in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who have received a diagnosis (not under evaluation) of PTSD and/or ADHD
* Understanding English or Swedish languages.

Exclusion Criteria:

* Ongoing substance use,
* active manic periods,
* psychotic disorders,
* suicidality,
* cognitive impairment.
* serious physical illness prohibiting participation in physical activities.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative experience score CPSS-5-S | 8 weeks
  Child PTSD Symptom Scale: 27-item self-report version rates each item from 0 (not at all) to 4 (6 or more times a week/almost always) based on the frequency and severity of the reported symptom experienced during the last month. The total severity score ranges from 0 to 80 and is calculated by summing the ratings of the first 20 items.
  The CPSS-5 also yields subscale scores for intrusion (Items 1-5), avoidance (Items 6-7), changes in cognition and mood (Items 8-14), and increased arousal and reactivity (Items15-20). Finally, seven items assess impairment of endorsed symptoms on daily functioning pertinent to youth (e.g., fun things you want to do, doing your chores, relationships with your friends). The respondent rates these items on a scale of 0 (not at all) to 4 (6 or more times a week/almost always), resulting in an impairment score that ranges from 0 to 28.
Inattention, impulsivity score | 8 weeks
  Parent-rated ADHD score, SNAP-IV: The SNAP-IV consists of a total of 26 questions, divided into two subscales: one for inattention symptoms and one for hyperactivity-impulsivity symptoms. Each subscale contains 9 items, and there are 8 additional questions that provide an overall assessment of impairment. Higher score indicates higher problem load.
Resilience score | 8 weeks
  social, ecological, psychological, and emotional resilience: The Child and Youth Resilience Measure-Revised-Adapted Swedish (CYRM-R-AS) is a self-report measures of social ecological and psychological, emotional resilience. In addition to an overall score of resilience, scores can be derived for the three subscales of the measures personal, caregiver and psychological/emotional resilience. The CYRM-R (simplified) is suitable for youth aged 10-23 with difficulties to comprehend text or sustain attention. Its 23 items can be scored on 3- point Likert scales. The items in the measure are all positively worded and therefore scoring involves simple summing of responses. It can be used to evaluate the efficacy of interventions to build and maintain resilience. Three sub-scales can be created . Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Pain frequency and intensity | 8 weeks
  Pain frequency, intensity and location: The Pain assessment instrument uses verbal and numerical assessment scales, where the participant describes their pain during the last month using words (no pain; mild pain; moderate pain; severe pain; very severe pain; unbearable pain) and using numbers between 0 and 10, where 0 (zero) represents no pain, and 10 represents the worst possible pain. Primary and secondary pain localization is described in free text by the participant. Higher scores indicate increased problem load
affect | 8 weeks
  Positive and Negative affect state: The Positive Affect and Negative Affect-Extended (PANAS-X) instrument consists of 30 items and captures the valence (positive and negative) and the arousal (high or low) of the mood descriptors during the last month.
  The following are examples for all four categories. Positive activated: active, enthusiastic, excited, inspired, and proud; Positive deactivated: at ease, serene, calm, relaxed, and content; Negative activated: afraid, scared, hostile, guilty, and ashamed; Negative deactivated: tired, sluggish, drowsy, dull, and bored.
  HIgher scores indicate dominance of the specific subscale in affect state.
Self-directednes | 8 weeks
  Self-control, responsibility: Self-Directedness character domain of the J-TCI (Junior Temperament and Character Inventory, Cloninger et al., Swedish version: Kerekes et al.) has been used to measure changes in this domain during the last month. Has been used for 9-15-year-old adolescents in Sweden. Self-directedness, or self-determination, refers to a tendency to achieve personal goals and values. Includes 20 questions and dichotomic responses (Yes/No). Higher scores indicate better outcome.
Quality of life score | 8 weeks
  PedsQL and PedsQL FIM: The 23-item PedsQL™ 4.0 Generic Core Scales encompass:
  * 1) Physical Functioning (8 items),
  * 2) Emotional Functioning (5 items),
  * 3) Social Functioning (5 items), and
  * 4) School Functioning (5 items), and were developed through focus groups, cognitive interviews, pre-testing, and field-testing measurement development protocols.
  The Parent-reported Health-Related Quality of Life of the Child (PedsQL-Fam) inventory is an assessment tool designed to measure the health-related quality of life (HRQOL) of children from the perspective of their parents or caregivers. It includes questions about different aspects of the child's functioning and well-being, 25 items. Higher scores indicate better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Sylvia Child Hospital , CAP, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of data collection and analyses, and after we coudl publish the results in peer reviewed scientific journals

REFERENCES:
- See also: The project's home page that includes this study as well. — https://www.yogatocare.com/